CLINICAL TRIAL: NCT03339219
Title: A Phase 2, Open-Label, Single-Arm Study of Cabozantinib in Japanese Patients With Advanced Renal Cell Carcinoma That Has Progressed After Prior VEGFR Tyrosine Kinase Inhibitor Therapy
Brief Title: A Phase 2 Study of Cabozantinib in Japanese Participants With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cabozantinib-2001; U1111-1201-4230 (Other: WHO); JapicCTI-173763 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Results first posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Advanced Renal Cell Carcinoma
Keywords: Drug Therapy
MeSH Terms: interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib 60 mg (Experimental): Cabozantinib 60 mg, tablet, orally, once daily (QD) in the fasted state until unacceptable toxicity or need for subsequent systemic anticancer treatment up to 2.5 years.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib tablets
  Other Names: XL184

SUMMARY:
The purpose of this study is to evaluate the efficacy of cabozantinib measured by Independent Radiology Committee (IRC)-assessed objective response rate (ORR) in Japanese participants with advanced renal cell carcinoma (RCC) that has progressed after prior vascular endothelial growth factor receptor (VEGFR) tyrosine kinase inhibitor (TKI) therapy.

DETAILED DESCRIPTION:
The drug being tested in this study is called cabozantinib. Cabozantinib is being tested to treat people who have advanced renal cell carcinoma. This study will look at the efficacy of cabozantinib.

The study will enroll approximately 35 patients. Participants will be enrolled in one treatment group in non-randomized and opened manner:

• Cabozantinib 60 mg

All participants will be asked to take tablets of cabozantinib at once daily in the fasted state throughout the study.

This multi-center trial will be conducted in Japan. The overall time to participate in this study is approximately at most 3 years. Participants will make multiple visits to the clinic in treatment period, and posttreatment period including a follow-up assessment after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Japanese participants 20 years of age or older on the day of consent.
* Documented histological or cytological diagnosis of renal cell carcinoma (RCC) with a clear-cell component.
* Measurable disease per RECIST 1.1 as determined by the investigator.
* Must have received at least one VEGFR-targeting TKI (eg, sorafenib, sunitinib, axitinib, pazopanib or tivozanib).
* For the most recently received VEGFR-targeting TKI the following criteria must apply:

  * Must have radiographically progressed during treatment, or been treated for at least 4 weeks and radiographically progressed within 6 months after the last dose.

Radiographic progression is defined as unequivocal progression of existing tumor lesions or developing new tumor lesions as assessed by the investigator on computerized tomography (CT) or magnetic resonance imaging (MRI) scans.

- The last dose must have been within 6 months before the first day of study drug administration (Week 1 Day 1).

* Recovery to baseline or ≤Grade 1 Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
* Karnofsky Performance Status (KPS) score of ≥70%.
* Adequate organ and marrow function at Screening.

Exclusion Criteria:

* Prior treatment with everolimus, or any other specific or selective target of rapamycin complex 1/phosphoinositide 3-kinase/AKT inhibitor (eg, temsirolimus), or cabozantinib.
* Receipt of any type of small-molecule kinase inhibitor (including investigational kinase inhibitor) within 14 days before Week 1 Day 1.
* Receipt of any type of anticancer antibody (including investigational antibody) within 28 days before Week 1 Day 1.
* Radiation therapy for bone metastasis within 14 days, and/or any other external radiation therapy within 28 days before Week 1 Day 1. Systemic treatment with radionuclides within 42 days before Week 1 Day 1.

Participants with clinically relevant ongoing complications from prior radiation therapy are not eligible.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (19):
- Japan (19):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kindai University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Nippon Medcal School Hospital, Bunkyo-ku, Tokyo
  - Toranomon Hospital, Minato-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Kyushu University Hospital, Fukuoka
  - Niigata University Medical and Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Osaka City University Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Tokushima University Hospital, Tokushima
  - Yamagata University Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Nakaigawa N, Tomita Y, Tamada S, Tatsugami K, Osawa T, Oya M, Kanayama H, Miura Y, Sassa N, Nishimura K, Nozawa M, Masumori N, Miyoshi Y, Kuroda S, Kimura A. Final efficacy and safety results and biomarker analysis of a phase 2 study of cabozantinib in Japanese patients with advanced renal cell carcinoma. Int J Clin Oncol. 2023 Mar;28(3):416-426. doi: 10.1007/s10147-022-02283-w. Epub 2023 Jan 3. PMID 36595123
- [Derived] Tomita Y, Tatsugami K, Nakaigawa N, Osawa T, Oya M, Kanayama H, Nakayama Kondoh C, Sassa N, Nishimura K, Nozawa M, Masumori N, Miyoshi Y, Kuroda S, Tanaka S, Kimura A, Tamada S. Cabozantinib in advanced renal cell carcinoma: A phase II, open-label, single-arm study of Japanese patients. Int J Urol. 2020 Nov;27(11):952-959. doi: 10.1111/iju.14329. Epub 2020 Aug 12. PMID 32789967

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 16 investigative sites in Japan from 13 December 2017 to 25 August 2020.
Pre-assignment Details: Participants with a diagnosis of advanced renal cell carcinoma (RCC) were enrolled in a single-arm study to receive cabozantinib 60 mg, tablet, orally, once daily.
Period: Overall Study
Arm/Group | Cabozantinib 60 mg
Started | 35
Completed | 0
Not Completed | 35
Not completed — Death | 12
Not completed — Site Terminated by Sponsor | 22
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least one dose of study drug.
Arm/Group | Cabozantinib 60 mg
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 35
Memorial Sloan-Kettering Cancer Center (MSKCC) Risk Factors [Count of Participants; unit: Participants] — MSKCC was used to determine the prognostic risk score in participants with advanced RCC. The risk factors for RCC were graded as 0 to 3, where 0=favorable, 1=intermediate, 2 or 3= poor.
  Participants
    Favorable Risk (0) | 11
    Intermediate Risk (1) | 19
    Poor Risk (2 or 3) | 5
Heng Criteria [Count of Participants; unit: Participants] — Heng criteria assess prognostic risk in RCC participants. The score ranges from 0 to 6, where 0 (favorable), 1-2 (intermediate), and 3-6 (poor).
  Participants
    Favorable Risk (0) | 6
    Intermediate Risk (1-2) | 22
    Poor Risk (3-6) | 7
Karnofsky Performance Status (PS) [Count of Participants; unit: Participants] — Karnofsky PS is used to quantify participant's general well-being and activities of daily life and participants are classified based on their functional impairment. Karnofsky PS score is 11 level score which ranges between 0 (dead) to 100 (normal, no complaints, no evidence of disease). Higher score means higher ability to perform daily tasks. Only categories with participants are reported.
  Participants
    70 (Cares for self, unable to carry on normal activity or to do active work) | 1
    80 (Normal activity with effort; some signs or symptoms of disease) | 5
    90 (Able to carry on normal activity; minor signs or symptoms of disease) | 5
    100 (Normal, no complaints, no evidence of disease) | 24
Eastern Cooperative Oncology (ECOG) Group PS [Count of Participants; unit: Participants] — The ECOG scale assess participant's ability to perform daily activities as:Grade 0:fully active,able to carry on pre-disease activities without restriction;Grade 1:restricted in physically strenuous activity,but ambulatory,able to carry work of light or sedentary nature;Grade 2:ambulatory,capable of all self-care but unable to carry out any work activities;Grade 3:capable of only limited self-care,confined to bed or chair >50% of waking hours;Grade 4:completely disabled.Cannot carry on any self-care,totally confined to bed or chair;Grade 5:death.Only categories with participants are reported.
  Participants
    Grade 0 | 26
    Grade 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants whose best overall response was complete response (CR) or partial response (PR) evaluated by the independent review committee (IRC) per response evaluation criteria in solid tumors version 1.1 (RECIST V1.1) which was confirmed by a subsequent evaluation conducted ≥28 days later. Per RECIST V1.1, CR was defined as the disappearance of all lesions, and all pathological lymph nodes (whether target or nontarget) must have a reduction in short axis to <10 millimeter (mm). PR was defined as at least a 30% decrease in the sum of diameter (SoD) of target lesions, taking as a reference the Baseline SoD.
Time Frame: From first dose of study drug up to first documentation of CR or PR (up to 2.5 years)
Population: FAS included all participants who received at least one dose of study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib 60 mg
Number analyzed (Participants) | 35
percentage of participants | 25.7 [14.122 to 40.582]

2. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as percentage of participants whose best overall response is CR, PR, or stable disease (SD) per RECIST V1.1. Response and progression were evaluated by IRC per RECIST V1.1. CR and PR required confirmation by a subsequent evaluation conducted ≥28 days later and an assessment of SD was made at least 8 weeks after the first day of study drug. Per RECIST V1.1, CR was defined as the disappearance of all lesions, and all pathological lymph nodes (whether target or nontarget) must have a reduction in the short axis to <10 mm. PR was defined as at least a 30% decrease in SoD of target lesions, taking as a reference the Baseline SoD. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: From first dose of study drug up to first documentation of CR or PR or SD (up to 2.5 years)
Population: FAS included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib 60 mg
Number analyzed (Participants) | 35
percentage of participants | 85.7 [69.743 to 95.194]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the first day of study drug administration to the earlier of progressive disease (PD) per RECIST V1.1 or death due to any cause. Per RECIST V1.1, PD was defined at least a 20% increase in the SoD of target lesions, taking as a reference the smallest (nadir) SoD since (and including) Baseline. In addition to the relative increase of 20%, the SoD also demonstrated an absolute increase of at least 5 mm.
Time Frame: From first dose of study drug up to disease progression or death (up to 2.5 years)
Population: FAS included all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib 60 mg
Number analyzed (Participants) | 35
months | 11.1 [7.4 to 18.4]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the first day of study drug administration to death due to any cause.
Time Frame: From first dose of study drug up to death due to any cause (up to 2.5 years)
Population: FAS included all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib 60 mg
Number analyzed (Participants) | 35
months | NA [23.4 to NA] — Median and upper limit for 95% confidence interval (CI) was not estimable due to the low number of participants with events.

5. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. TEAEs were defined as AEs whose date of onset occurs on or after the start of study drug and within 30 days after the last dose of study treatment.
Time Frame: From first dose up to 30 days after the last dose of the study drug (up to 2.6 years)
Population: Safety Analysis Set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cabozantinib 60 mg
Number analyzed (Participants) | 35
percentage of participants | 100.0

6. Secondary Outcome: Percentage of Participants With Grade 3 or Higher TEAEs
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. TEAEs were defined as AEs whose date of onset occurs on or after the start of study drug and within 30 days after the last dose of study treatment. Severity grade was defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. As per the NCI-CTCAE, Grade 1 scales as mild; Grade 2 scales as moderate; Grade 3 scales as severe or medically significant but not immediately life-threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to AE.
Time Frame: From first dose up to 30 days after the last dose of the study drug (up to 2.6 years)
Population: Safety Analysis Set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cabozantinib 60 mg
Number analyzed (Participants) | 35
percentage of participants | 82.9

7. Secondary Outcome: Percentage of Participants With Serious TEAEs
Description: A serious TEAE was any untoward medical occurrence or effect that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was medically important due to other reasons than the above-mentioned criteria. TEAEs were defined as AEs whose date of onset occurs on or after the start of study drug and within 30 days after the last dose of study treatment.
Time Frame: From first dose up to 30 days after the last dose of the study drug (up to 2.6 years)
Population: Safety Analysis Set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cabozantinib 60 mg
Number analyzed (Participants) | 35
percentage of participants | 42.9

8. Secondary Outcome: Percentage of Participants With TEAEs Leading to Permanent Treatment Discontinuation
Description: as for outcome 5
Time Frame: From first dose up to 30 days after the last dose of the study drug (up to 2.6 years)
Population: Safety Analysis Set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cabozantinib 60 mg
Number analyzed (Participants) | 35
percentage of participants | 17.1

9. Secondary Outcome: Percentage of Participants With TEAEs Leading to Dose Modification (Dose Reduction or Interruption)
Description: as for outcome 5
Time Frame: From first dose up to 30 days after the last dose of the study drug (up to 2.6 years)
Population: Safety Analysis Set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cabozantinib 60 mg
Number analyzed (Participants) | 35
percentage of participants
  Dose Reduction | 88.6
  Dose Interruption | 80.0

10. Secondary Outcome: Percentage of Participants With Clinically Significant Abnormal Laboratory Values
Description: Clinical laboratory tests included tests of serum chemistry, hematology, urine chemistry, coagulation, and thyroid function prespecified in the protocol. Only those categories are reported which are considered clinically significant abnormal laboratory values post baseline, as assessed by the investigator.
Time Frame: From first dose up to 30 days after the last dose of the study drug (up to 2.6 years)
Population: Safety Analysis Set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cabozantinib 60 mg
Number analyzed (Participants) | 35
percentage of participants
  White Blood Cells (WBC) Decreased | 17.1
  Absolute Neutrophil Count (ANC) Decreased | 5.7
  Lymphocytes Increased | 2.9
  Lymphocytes Decreased | 34.3
  Platelets Decreased | 20.0
  Hemoglobin Increased | 2.9
  Hemoglobin Decreased | 85.7
  Albumin Decreased | 88.6
  Alkaline Phosphatase (ALP) Increased | 65.7
  Amylase Increased | 57.1
  Alkaline Phosphatase (ALT) Increased | 74.3
  Aspartate Aminotransferase (AST) Increased | 80.0
  Corrected Calcium Increased | 5.7
  Corrected Calcium Decreased | 8.6
  Creatinine Increased | 97.1
  Gamma-glutamyl Transferase (GGT) Increased | 54.3
  Glucose Increased | 62.9
  Glucose Decreased | 5.7
  Lactate Dehydrogenase (LDH) Increased | 100
  Lipase Increased | 45.7
  Magnesium Increased | 14.3
  Magnesium Decreased | 77.1
  Phosphate Decreased | 54.3
  Potassium Increased | 14.3
  Potassium Decreased | 22.9
  Sodium Decreased | 48.6
  Total Bilirubin Increased | 17.1
  Urine Protein-to-creatinine Ratio (UPCR) Increased | 91.4

11. Secondary Outcome: Percentage of Participants With Clinically Significant Abnormal Vital Sign
Description: Vital signs included diastolic blood pressure (DBP) and systolic blood pressure (SBP) in the sitting position, pulse rate respiratory rate temperature, and weight. Abnormal vital sign values considered by the investigator to be clinically significant are reported as categories.
Time Frame: From first dose up to 30 days after the last dose of the study drug (up to 2.6 years)
Population: Safety Analysis Set included all participants who received at least one dose of study drug. Number analyzed are the number of participants with data available for analyses in the given category.
Measure: Number; unit: percentage of participants
Arm/Group | Cabozantinib 60 mg
Number analyzed (Participants) | 35
percentage of participants
  BP Increased: SBP <120 millimeters of mercury (mmHg) and DBP <80 mmHg: number analyzed (Participants) | 34
  BP Increased: SBP <120 millimeters of mercury (mmHg) and DBP <80 mmHg | 2.9
  BP Increased: SBP 120<= - <=139 mmHg or DBP 80<= - <=89 mmHg: number analyzed (Participants) | 34
  BP Increased: SBP 120<= - <=139 mmHg or DBP 80<= - <=89 mmHg | 11.8
  BP Increased: SBP 140<= - <=159 mmHg or DBP 90<= - <=99 mmHg: number analyzed (Participants) | 34
  BP Increased: SBP 140<= - <=159 mmHg or DBP 90<= - <=99 mmHg | 64.7
  BP Increased: SBP 160 mmHg<= and DBP <120 mmHg, or DBP 100<=- <=119 mmHg: number analyzed (Participants) | 34
  BP Increased: SBP 160 mmHg<= and DBP <120 mmHg, or DBP 100<=- <=119 mmHg | 20.6
  Weight Decreased >=10% from Baseline | 37.1

ADVERSE EVENTS:
Time Frame: Up to 2.6 years
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cabozantinib 60 mg
All-Cause Mortality (participants affected / at risk) | 12/35
Serious Adverse Events (participants affected / at risk) | 15/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib 60 mg (N=35)
Ileus (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Amylase increased (Investigations) | 1
Lipase increased (Investigations) | 1
Pancreatic enzymes increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain oedema (Nervous system disorders) | 1
Spinal cord disorder (Nervous system disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib 60 mg (N=35)
Anaemia (Blood and lymphatic system disorders) | 6
Hypothyroidism (Endocrine disorders) | 6
Cataract (Eye disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 24
Stomatitis (Gastrointestinal disorders) | 15
Constipation (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 6
Dental caries (Gastrointestinal disorders) | 4
Periodontal disease (Gastrointestinal disorders) | 4
Toothache (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Malaise (General disorders) | 11
Pyrexia (General disorders) | 8
Fatigue (General disorders) | 6
Oedema peripheral (General disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 13
Hepatobiliary disease (Hepatobiliary disorders) | 2
Contrast media allergy (Immune system disorders) | 2
Nasopharyngitis (Infections and infestations) | 8
Gingivitis (Infections and infestations) | 4
Periodontitis (Infections and infestations) | 3
Angular cheilitis (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 2
Skin infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Tooth fracture (Injury, poisoning and procedural complications) | 3
Limb injury (Injury, poisoning and procedural complications) | 2
Weight decreased (Investigations) | 14
Aspartate aminotransferase increased (Investigations) | 9
Alanine aminotransferase increased (Investigations) | 7
Blood thyroid stimulating hormone increased (Investigations) | 5
Amylase increased (Investigations) | 4
Blood alkaline phosphatase increased (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 3
Blood creatinine increased (Investigations) | 2
Blood lactate dehydrogenase abnormal (Investigations) | 2
Lipase increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Dysgeusia (Nervous system disorders) | 15
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 5
Proteinuria (Renal and urinary disorders) | 17
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 23
Rash (Skin and subcutaneous tissue disorders) | 7
Hair colour changes (Skin and subcutaneous tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT03339219/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT03339219/SAP_001.pdf